CLINICAL TRIAL: NCT02885428
Title: Silent Myocardial Ischemia in Patients With Diabetes Type 2: Diagnostic Value of Myocardial Strains Left Ventricular Resting Echocardiography 2D and 3D, Compared to Stress Echocardiography
Brief Title: Detection no Invasive of a Silent Myocardial Ischemia
Status: Terminated | Type: Observational
Why Stopped: Difficulties in the inclusion of patients with cardiacly asymptomatic type 2 diabetes and with at least two cardiovascular risk factors.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01458-39
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Silent Myocardial Ischemia; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: echography

SUMMARY:
The pathophysiological features of myocardial diabetic subject combined with cardiac autonomic neuropathy were behind the quietness of myocardial ischemia, known as silent myocardial ischemia (IMS). These patients have the risk to remain asymptomatic until the sudden onset of a myocardial infarction, or even sudden death.

That is why the investigators want to evaluate the contribution of non-invasive tools to stand in the diagnosis of IMS patients with diabetes type 2, asymptomatic heart on map: Technical myocardial speckle tracking in studying strains overall average left ventricular (longitudinal, circumferential and radial) measured in 2D and 3D at rest, compared to stress echocardiography with dobutamine (ESD)

ELIGIBILITY:
Inclusion Criteria:

* With at least two cardiovascular risk factors including: hypertension, dyslipidemia, smoking active or interrupted for less than 3 years, family history (relatives of the 1st degree) Accident major CV before 60.
* Or whatever the level of risk factors: peripheral artery disease and / or carotid atherosclerosis, or proteinuria

Exclusion Criteria:

* Valvular heart disease (severe to moderate valvular ) , hypertrophic , dilated , chronic lung
* History of cardiotoxic chemotherapy
* Atrioventricular blocks of degree
* Asthma
* Recent stroke within a month
* Bilateral carotid stenosis tight
* Glaucoma untreated narrow angle
* Subject to exclusion period (determined by a previous study or in progress)
* Inability to give informed about information
* patient under judicial protection
* patient guardianship or curatorship
* Current pregnancy (women of childbearing age )
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes, men or women, asymptomatic on the heart level, high risk
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
diagnostic of the silent myocardial ischemia | 80 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Samy TALHA, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No